CLINICAL TRIAL: NCT01156103
Title: Reducing Pediatric Obesity Through After-school Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Unified School District (Unknown); America SCORES, Bay Area (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H48814-32411-0; 1K23HD054470-01A1 (NIH)
Record Dates: First submitted 2009-02-17; First posted 2010-07-02 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
Keywords: obesity; minority; child; physical fitness; school; physical activity
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCORES (Experimental): America SCORES, Bay Area, after-school program
  Interventions: Behavioral: America SCORES, Bay Area
- Usual care (No Intervention): Standard after-school programming

INTERVENTIONS:
Behavioral: America SCORES, Bay Area — After-school program promoting physical activity via soccer 3 days/week
  Arms: SCORES

SUMMARY:
This study will assess the impact of a national, community-based after-school program promoting physical activity (America SCORES) on obesity, fitness and important cardiovascular risk factors among minority children. The investigators central hypothesis is that established community-based programs, such as America SCORES, can reduce obesity and cardiovascular risk among participants. The 1-year study followed 158 children from 6 public schools, 3 of which were randomized to have SCORES and 3 to "usual care" after-school program. Primary outcomes are change in body mass index (BMI), physical activity (measured by accelerometer), and fitness (aerobic capacity assessed with the 20-meter shuttle test). Cardiovascular outcomes include blood pressure, body composition (assessed using bioelectrical impedance) and waist circumference. The investigators will also measure academic outcomes.

DETAILED DESCRIPTION:
Baseline measures were collected in September 2009; midpoint measures were collected in January 2010; and final measures were collected in May 2010. Repeated measures analyses will compare trajectories for BMI, physical activity, and fitness between students in the SCORES and the usual care arms.

ELIGIBILITY:
Inclusion Criteria:

* 3rd-5th grade student enrolled in after-school program in San Francisco Unified School District

Exclusion Criteria:

* Uncontrolled asthma
* Unable to participate in moderate physical activity

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in BMI z-score | Baseline (0 months) and 9 months

SECONDARY OUTCOMES:
Change in Aerobic capacity | Baseline and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Kristine A Madsen, MD, MPH, Principal Investigator — University of California, San Francisco

REFERENCES:
- [Derived] Madsen K, Thompson H, Adkins A, Crawford Y. School-community partnerships: a cluster-randomized trial of an after-school soccer program. JAMA Pediatr. 2013 Apr;167(4):321-6. doi: 10.1001/jamapediatrics.2013.1071. PMID 23440308